CLINICAL TRIAL: NCT00099099
Title: Dietary Energy Restriction and Metabolic Aging in Humans
Brief Title: CALERIE (Tufts) - Comprehensive Assessment of Long-term Effects of Reducing Intake of Energy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute on Aging (NIA) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AG0006; 3U01AG020480 (NIH)
Record Dates: First submitted 2004-12-08; First posted 2004-12-09 (Estimated); Last update posted 2009-12-11 (Estimated); Status verified 2006-02

CONDITIONS: Aging
Keywords: Longevity; Calorie restriction; Physical activity; Weight loss
MeSH Terms: conditions — Motor Activity; Weight Loss | interventions — Caloric Restriction

INTERVENTIONS:
Behavioral: Caloric Restriction (CR)

SUMMARY:
This study is one of three CALERIE trials that test the hypothesis that a reduced calorie, nutritionally sound diet increases the length of life and prevents some age-related chronic diseases such as cancer, diabetes, and cardiovascular disease. The three sites that are participating in the CALERIE trial represent a diversity of subject populations and interventional strategies.

DETAILED DESCRIPTION:
Researchers at the Jean Mayer USDA Human Nutrition Research Center on Aging at Tufts University are enrolling overweight men and women aged 20-42 in a 1-year study to develop an effective calorie restricted regimen that minimizes hunger and prevents weight regain. The study also examines the effects of weight loss on body composition, metabolism and aging. Two different diets containing usual foods and a healthy balance of nutrients will be tested at 2 levels of caloric restriction, 10% and 30% (in other words, 90% or 70% of what one would normally eat). Weight loss is expected for most volunteers participating in this study, but cannot be guaranteed.

ELIGIBILITY:
Inclusion Criteria

* Healthy men and women
* Body mass index (BMI) = 25-30
* Slightly overweight, < 275 lbs
* Women 25-45, pre-menopause
* Men 25-50
* Not traveling often or planning to move

Exclusions:

* Cardiovascular disease or blood pressure greater than 160/90
* Diabetes
* Major psychiatric disorders
* Eating disorders
* Post obese; previous BMI > 32
* Weight change of more than ten pounds in the past 90 days
* Over 275 pounds
* Smoking
* Regular exercise, more than twice per week
* Current prescription drug use, except oral contraceptives
* Alcoholism or substance abuse
* Pregnant or lactating (breast feeding), planning to become pregnant, or not regularly using contraception
* Abnormal electrocardiogram (EKG)
* Local resident for less than one year
* Occupations requiring full alertness and motor skills, with no allowance for a chance of postural dizziness (airline pilots, etc.)
* Injuries by any metallic object that is still present in the body
* Braces, non-removable dentures, or non-removable bridgework

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44
Dates: Start 2002-03; Primary Completion 2004-12 (Actual); Study Completion 2004-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan B. Roberts, PhD, Principal Investigator — Jean Mayer USDA HNRCA at Tufts University
Locations (1):
- Jean Mayer USDA Human Nutrition Research Center on Aging at Tufts University, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Karl JP, Cheatham RA, Das SK, Hyatt RR, Gilhooly CH, Pittas AG, Lieberman HR, Lerner D, Roberts SB, Saltzman E. Effect of glycemic load on eating behavior self-efficacy during weight loss. Appetite. 2014 Sep;80:204-11. doi: 10.1016/j.appet.2014.05.017. Epub 2014 May 21. PMID 24859114
- [Derived] Racette SB, Das SK, Bhapkar M, Hadley EC, Roberts SB, Ravussin E, Pieper C, DeLany JP, Kraus WE, Rochon J, Redman LM; CALERIE Study Group. Approaches for quantifying energy intake and %calorie restriction during calorie restriction interventions in humans: the multicenter CALERIE study. Am J Physiol Endocrinol Metab. 2012 Feb 15;302(4):E441-8. doi: 10.1152/ajpendo.00290.2011. Epub 2011 Nov 29. PMID 22127229